CLINICAL TRIAL: NCT06658951
Title: Exploratory Study to Evaluate the Safety and Preliminary Efficacy of Anti-HER2 CAR-T Cell Injection in Patients With HER2-positive Advanced Malignant Solid Tumors
Brief Title: Anti-HER2 CAR-T Cell Injection in Patients With HER2-positive Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UTC Therapeutics Inc. (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anti-HER2 CAR-T
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-10

CONDITIONS: HER2-positive Advanced Malignant Solid Tumors
Keywords: Anti-HER2 CAR-T; Solid tumor

STUDY DESIGN:
Intervention Model Description: Accelerated titration and 3+3 design dose escalation phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-HER2 CAR-T cells (Experimental): All eligible participants will receive a conditioning chemotherapy regimen of fludarabine, cyclophosphamide and ABRAXANE followed by Anti-HER2 CAR-T cell injection.
  Interventions: Biological: Anti-HER2 CAR-T cells

INTERVENTIONS:
Biological: Anti-HER2 CAR-T cells — All eligible participants will receive a conditioning chemotherapy regimen of fludarabine, cyclophosphamide and ABRAXANE followed by Anti-HER2 CAR-T cell injection.

SUMMARY:
This is a single-arm, open-label, exploratory clinical study to evaluate the safety and preliminary efficacy of Anti-HER2 CAR-T cell injection in patients with HER2-positive advanced malignant solid tumors.

DETAILED DESCRIPTION:
All eligible participants will receive a conditioning chemotherapy regimen of fludarabine, cyclophosphamide and ABRAXANE followed by Anti-HER2 CAR-T cell injection.The dose escalation phase will determine the maximum tolerated dose (MTD) of Anti-HER2 CAR-T cell injection. Additional patients will be enrolled in the dose expansion phase to further characterize the safety profile and evaluate the efficacy of Anti-HER2 CAR-T cell injection, and establish recommended phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 to 70 years old (including cut-off value), gender is not limited.

  2. Solid tumors that histological diagnosis of malignancy refractory to, or relapsing after standard therapy, including but not limited to gastric cancer, biliary system tumors, bladder cancer, ovarian cancer, endometrial cancer, cervical cancer, colorectal cancer, breast cancer, lung cancer, esophageal cancer, etc.

  3. At least one measurable lesion according to RECIST v1.1.

  4. HER2 should be positive confirmed by Immunohistochemistry in tumor tissue samples.

  5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

  6. Life expectancy ≥ 3 months.

  7. The organ function must meet the protocol requirements.

  8. Female participants of childbearing potential must undergo a pregnancy test and the results must be negative. Female participants of childbearing potential or male participants whose sex partner has childbearing potential must be willing to use effective methods of contraception from screening period to at least 1 year after infusion.

  9. Participants must be able to understand the protocol and be willing to enroll the study, sign the informed consent, and be able to comply with the study and follow-up procedures.

Exclusion Criteria:

* 1. Pregnant or lactating women.

  2. Patients with hepatitis B surface antigen (HBsAg) positive. Patients who is hepatitis B core antibody (HBcAb) positive and the quantification of HBV DNA in peripheral blood is higher than the lower limit of detection. Patients who is hepatitis C virus (HCV) antibody positive and quantification of HCV DNA in peripheral blood is higher than the lower limit of detection. Patients with human immunodeficiency virus (HIV) antibody positive, or syphilis antibody positive.

  3. The toxicities caused by the prior therapy (surgery, chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.) have not recovered to grade 1 according to CTCAE, except for hair loss and peripheral sensory nerve disorders.

  4. Have received any allogeneic tissue/organ transplantation (including bone marrow transplantation, stem cell transplantation, liver transplantation, kidney transplantation), except for the transplantation that does not require immunosuppressive therapy (such as: corneal transplantation, hair transplantation.)

  5. Patients have received anti-HER2 CAR-T cell therapy.

  6. Patients who have history of major surgery and unrecovered severe trauma within 4 weeks prior to signing informed consent; or plan to have major surgery within 12 weeks of cell therapy.

  7. Presence of known central nervous system metastases, but the following patients will be allowed: a) Asymptomatic brain metastases; b) Clinically stable (no radiographic progression within 4 weeks before apheresis and return of any neurologic symptoms to baseline), and with no need for corticosteroids or other treatment for brain metastases for ≥ 4 weeks.

  8. Patients with clinically significant systemic disease (such as: severe active infection or significant cardiac, pulmonary, hepatic, nervous system, or other organ dysfunction) that evaluated by the investigator would impair the patients' ability to tolerate the treatments used in this study or significantly increase the risk of complications.

  9. History of severe systemic hypersensitivity reaction to the drugs/ingredients [fludarabine, cyclophosphamide, dimethyl sulfoxide (DMSO), low molecular dextran, human serum albumin (HSA), etc.] used in this study.

  10. Patients have received attenuated vaccine within 4 weeks prior to signing informed consent.

  11. Patients have received other clinical trials within 4 weeks prior to signing informed consent.

  12. History of another malignancy tumor within the previous five years, except for adequately treated non-melanoma skin cancer, carcinoma in situ of bladder, stomach, colon, cervix/dysplasia, melanoma, or breast.

  13. History of neuropsychiatric diseases diagnosed by the ICD-11 criteria or evaluated by investigator, including but not limited to epilepsy, schizophrenia, dementia, drug and alcohol addictions.

  14. For any other reasons, the patients are believed not suitable for participation in this study by investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Identification of Maximum Tolerated Dose (MTD) & Incidence of Dose-limiting Toxicities (DLTs) | 4 weeks after the CAR-T cells infusion
  Incidence and severity of dose-limiting toxicities (DLTs) following infusion of CAR-T cell injection, at each dose level tested in dose escalation phase.
Adverse Events (AEs) | 2 years
  Incidence and severity of adverse events.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  The Objective Response Rate (ORR) is the percentage of participants who achieved Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1.
Disease Control Rate (DCR) | 2 years
  Disease control rate (DCR) is the percentage of participants who achieved Complete Response (CR) or Partial Response (PR) or Stable disease (SD) based on RECIST version 1.1.
Progression-Free Survival (PFS) | 2 years
  PFS is defined as the time from CAR-T infusion to the date of the disease progression or death from any cause.
Overall Survival (OS) | 2 years
  OS is defined as the time from CAR-T infusion to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No